CLINICAL TRIAL: NCT04997538
Title: Study on Susceptibility Genes of Anterior Cruciate Ligament, Patella Dislocation and Discoid Meniscus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2018245
Record Dates: First submitted 2021-06-25; First posted 2021-08-09 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-01

CONDITIONS: Gene Abnormality; Meniscus Injury; Cruciate Ligament Rupture
Keywords: gene; exon; cruciate ligament; patellar; meniscus injury
MeSH Terms: conditions — Patella Fracture

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Genomes of all sports medicine-related genes will be exome sequenced to find relevant gene mutations. To further study the molecular mechanisms and signaling pathways related to sports injury. To search for genetic risk factors of injury and put forward related scientific hypotheses. To demonstrate the importance of mutation or polymorphism of related genes in injury.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with joint sports injuries.
2. Follow-up patients after sports injury.
3. Patients with genetic predisposition to sports injuries.
4. Patients with family genetic predisposition to exercise-related diseases and their relatives.

Exclusion Criteria:

1. Patients with joint damage caused by external force.
2. The patient is accompanied by other injuries at the same time.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ACL injury surgery, patients after sports injury, knee joint shape abnormality, and patients with family genetic predisposition to sports related diseases
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Magnetic resonance imaging (MRI) | Before the operation
  All MRI scans were obtained with a 3.0-T MRI scanner (Magnetom Trio with TIM system, Siemens Healthcare). Five routine MRI sequences with a section thickness of 4 mm were obtained in all patients. Preoperative and postoperative evaluations of the articular cartilage of the transplanted compartment were performed with the Yulish score41 (grade 0 = normal; grade 1 = normal contour 6 abnormal signal; grade 2 = superficial fraying, erosion, or ulceration of <50%; grade 3 = partial-thickness defect of >50% but <100%; grade 4 = full-thickness cartilage loss). The signal of the meniscus allograft in the coronal plane of the T2-weighted fast spin echo sequence was graded on a scale of 0 to 3.
Magnetic resonance imaging (MRI) | an average of 1 year
  All MRI scans were obtained with a 3.0-T MRI scanner (Magnetom Trio with TIM system, Siemens Healthcare). Five routine MRI sequences with a section thickness of 4 mm were obtained in all patients. Preoperative and postoperative evaluations of the articular cartilage of the transplanted compartment were performed with the Yulish score41 (grade 0 = normal; grade 1 = normal contour 6 abnormal signal; grade 2 = superficial fraying, erosion, or ulceration of <50%; grade 3 = partial-thickness defect of >50% but <100%; grade 4 = full-thickness cartilage loss). The signal of the meniscus allograft in the coronal plane of the T2-weighted fast spin echo sequence was graded on a scale of 0 to 3.
Radiographs | Before the operation
  All patients also obtained 45° flexion weightbearing AP radiographs of both the ipsilateral and contralateral sides at final follow-up. The radiograph of the total length of the lower limbs was used to evaluate alignment. In the AP plain radiographs, the shortest distance between the femoral condyle and tibial plateau of the transplanted side was measured and designated as the joint space height. The difference between the ipsilateral and contralateral sides was calculated to identify joint space narrowing. In addition, Kellgren-Lawrence (K-L) grading was used to assess the osteoarthritic status of the knee.
Radiographs | an average of 1 year
  All patients also obtained 45° flexion weightbearing AP radiographs of both the ipsilateral and contralateral sides at final follow-up. The radiograph of the total length of the lower limbs was used to evaluate alignment. In the AP plain radiographs, the shortest distance between the femoral condyle and tibial plateau of the transplanted side was measured and designated as the joint space height. The difference between the ipsilateral and contralateral sides was calculated to identify joint space narrowing. In addition, Kellgren-Lawrence (K-L) grading was used to assess the osteoarthritic status of the knee.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lin, Study Director — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China